CLINICAL TRIAL: NCT03697772
Title: Continuity of Care and Use of Urgent Healthcare in Multimorbid Patients
Acronym: MULTIPASS-2
Status: Completed | Type: Observational
Sponsor: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, Alexandre MALMARTEL, Academic doctor of medicine, University of Paris 5 - Rene Descartes
Other Study IDs: 2018-A01159-46
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Multimorbidity; Continuity of Care
Keywords: continuity of care; primary care; multimorbidity; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multmorbid patients: patients with 2 chronic diseases (medical conditions requiring management for more than 6 months)

SUMMARY:
Chronic disease management is a public health problem that faces monitoring difficulties related to complex care pathways. This study will analyze the use of unscheduled or urgent care according to the continuity of care in multimorbid patients

DETAILED DESCRIPTION:
The prevalence of chronic diseases in the population is increasing significantly. It represents a new challenge for doctors and health authorities. However, patients often have at least two chronic diseases. These are referred to as "multimorbid" patients, whose continuity of care has not been well studied to date.

This observational study evaluates the association between the continuity of care in multimorbid patients seen in general practice and their use of urgent healthcare, their quality of life and their burden of treatment.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age, seen in consultation in the office by an investigating doctor, with a follow-up for more than 12 months in the office, presenting at least two chronic disease , having given their written consent to participate in the study

Exclusion Criteria:

* seen at home
* unable to respond (cognitive problems or language barrier)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: multimorbid primary care patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Continuity of care | over the past 1year
  Bice-Boxerman index, measuring continuity of care (from 0 to 1, 1 = good continuity of care)
care pathway | over the past 1 year
  the number of health care consultations with any physician (primary care, emergency department, hospitalisation), collected from the French national health insurance database

SECONDARY OUTCOMES:
global quality of life | over the past 1 year
  EuroQol Health Questionnaire in 5 questions measuring quality of life by the EuroQol Group. (from 0 to 100, 100= good quality of life)
burden of traitement | over the past 1 year
  Treatment Burden Questionnaire developped by VT Tran (from 0 to 130, 130 = treatments are a huge problem for the patient)

CONTACTS AND LOCATIONS:
Locations (1):
- Université Paris Cité, Paris, France

IPD SHARING:
Plan to Share IPD: No